CLINICAL TRIAL: NCT02703194
Title: A Study of Safety and Efficacy of Leflunomide for Maintenance of Remission in IgG4 Related Disease
Brief Title: Leflunomide for Maintenance of Remission in IgG4 Related Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhu, Deputy Director of Rheumatology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLAGH-IgG4
Record Dates: First submitted 2016-02-27; First posted 2016-03-09 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Immunoglobulin G4 Related Sclerosing Disease
Keywords: IgG4-related disease; IgG4-related sclerosing cholangitis; Mikulicz disease; Pancreatitis; Retroperitoneal fibrosis; Lymphadenopathy
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Mikulicz' Disease; Pancreatitis; Retroperitoneal Fibrosis; Lymphadenopathy | interventions — Prednisone; Prednisolone; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Prednisone mono-therapy
  Interventions: Drug: Prednisone
- Prednisone and Leflunomide (Experimental): Prednisone and Leflunomide combination therapy
  Interventions: Drug: Prednisone; Drug: Leflunomide

INTERVENTIONS:
Drug: Prednisone — Prednisone:A starting dose of 0. 5-0. 8mg/(kg*d) will be given. Following four-week period, the dose will be tapered gradually to 5mg/d until the end of 12 months of follow-up period.
  Other Names: Prednisolone
Drug: Leflunomide — Leflunomide:A starting dose of 20 mg/day will be given. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor adverse effects occur(e.g., liver enzyme elevations).
  Other Names: ARAVA®
  Arms: Prednisone and Leflunomide

SUMMARY:
The study has been designed as a 12-month, open-label, randomized, controlled study comparing the use of prednisone mono-therapy and prednisone and leflunomide combination therapy in treating patients with IgG4-related disease.

DETAILED DESCRIPTION:
The aim of this clinical trial is to determine the safety and efficacy of Leflunomide in treating patients with IgG4-related disease by comparing the outcomes of prednisone and leflunomide combination therapy with prednisone mono-therapy. The follow-up period will be 12 months. During the follow-up period, results of laboratory tests and image examinations, IgG4-RD RI and other parameters which can reflect treatment response as well as adverse effect events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Diagnosis of IgG4-RD according to either Consensus statement on the pathology of IgG4-related disease (for those who have undergone biopsies) or 2011 Comprehensive diagnostic criteria for IgG4-related disease. Both of the two criteria for diagnosis are specified below.

(1)Consensus statement on the pathology of IgG4-related disease

1. Histopathologic features consisting of dense lymphoplasmacytic infiltrate, fibrosis(usually storiform in character)and/or obliterative phlebitis within involved organs.
2. Either an elevated IgG4+/IgG+cell ratio of >40% within the affected organs or elevated IgG4-bearing plasma cells per high-power field is necessary. The cut-off number of IgG4-bearing plasma cells per high-power field is different depending upon the types of affected organs and specimens(through surgery or needle puncture biopsy).

(2)2011 Comprehensive diagnostic criteria for IgG4-related disease

1. Clinical examination showing characteristic diffuse/localized swelling or masses in single or multiple organs.
2. Hematological examination shows elevated serum IgG4 concentrations(135 mg/dl).
3. Histopathologic examination shows marked lymphocyte and plasmacyte infiltration and fibrosis or Infiltration of IgG4+ plasma cells(ratio of IgG4+/IgG+ cells > 40% and >10 IgG4+ plasma cells/HPF).

   Definite: a + b + c,Probable: a + c,Possible: a + b
4. Excluded from malignant tumors of each organ (e.g. cancer, lymphoma) and similar diseases (e.g. Sjögren's syndrome, primary sclerosing cholangitis, Castleman's disease, secondary retroperitoneal fibrosis, Wegener's granulomatosis, sarcoidosis, Churg-Strauss syndrome) by additional histopathological examination.
5. Even when patients cannot be diagnosed using the Comprehensive diagnostic criteria, they may be diagnosed using organ-specific diagnostic criteria for IgG4-RD, such as Diagnostic criteria for IgG4-Mikulicz's disease.

Exclusion Criteria:

1. Subjects having received steroids or immunosuppressants in recent 3 months will be excluded.
2. Subjects who were hypersensitive to leflunomide will be excluded.
3. ALT and/or AST is more than two folds of the upper limit of relevant reference value at baseline.
4. WBC is less than 3×10*9/L at baseline.
5. Female patients who are pregnant or breastfeeding.
6. Known significant concurrent medical disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Relapse rate at 12 months. | 12 months
  Relapse referred to the recurrence of previous clinical manifestations or abnormality of organ-specific imaging findings or serology tests after remission.

SECONDARY OUTCOMES:
Relapse rate at 6 months. | 6 months
  Relapse referred to the recurrence of previous clinical manifestations or abnormality of organ-specific imaging findings or serology tests after remission.
Complete response assessed by IgG4-RD Responder Index (IgG4-RD RI) at 1, 3, 6 and 12 months. | Up to 12 months
  Complete response (CR) is defined as IgG4-RD RI <3 at 1, 3, 6 and 12 months.
Partial response assessed by IgG4-RD RI at 1, 3, 6 and 12 months. | Up to 12 months
  Partial response (PR) is defined as IgG4-RD RI remaining ≥3 at 1, 3, 6 and 12 months.
Serum IgG4 concentrations (mg/dL) measured by immunonephelometry at 1, 3, 6 and 12 months. | Up to 12 months
Number of circulating plasmablasts (cell number/mL) assessed by flow cytometry by gating peripheral blood at 1, 3, 6 and 12 months. | Up to 12 months
Adverse effect events | Up to 12 months
  Treatment-related adverse effect, including abnormal liver function and leukopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Zhao Z, Gao D, Wang H, Liao S, Dong C, Luo G, Ji X, Li Y, Wang X, Zhao Y, Li K, Zhang J, Jin J, Zhang Y, Zhu J, Zhang J, Huang F. Additive effect of leflunomide and glucocorticoids compared with glucocorticoids monotherapy in preventing relapse of IgG4-related disease: A randomized clinical trial. Semin Arthritis Rheum. 2020 Dec;50(6):1513-1520. doi: 10.1016/j.semarthrit.2020.01.010. Epub 2020 Feb 3. PMID 32113839